CLINICAL TRIAL: NCT04990830
Title: Early Effects of Low Molecular Weight Heparin Therapy With Soft-Mist Inhaler for COVID-19 Induced Hypoxemia: A Phase IIb Trial
Brief Title: Effects of Low Molecular Weight Heparin Therapy With Soft-Mist Inhaler for COVID-19 Induced Hypoxemia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ayca Yildiz-Pekoz, Associate Professor, Istanbul University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-66175679-514.03.01-328141; 46325 (Other: Istanbul University Medical Faculty)
Record Dates: First submitted 2021-07-29; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome; Hypoxemia
Keywords: Heparin; Low Molecular Weight Heparin; Inhalation; Antiviral; Soft Mist Inhaler
MeSH Terms: conditions — Hypoxia; Respiratory Aspiration | interventions — enoxaparin sodium

STUDY DESIGN:
Intervention Model Description: Treatment Group - Control Group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhalation Treatment (Experimental): Treatment: Inhaled Low molecular weight heparin + Standard COVID-19 treatment,
  Inhaled Low molecular weight heparin (4000 IU given twice a day for 10 days)
  Interventions: Drug: Inhaled Low molecular weight heparin
- Control Group (Other): Treatment: Standard COVID-19 treatment
  Interventions: Drug: Standard Treatment

INTERVENTIONS:
Drug: Inhaled Low molecular weight heparin — Application with Soft Mist Inhaler
  Other Names: Enoxaparin Sodium
  Arms: Inhalation Treatment
Drug: Standard Treatment — Control Group
  Arms: Control Group

SUMMARY:
This is an investigator initiated, single-center, open-label, Phase IIb clinical trial with 40 patients (for a total of 80 patients) to assess efficacy of Low molecular weight heparin using soft mist inhaler in the treatment of critically ill patients with COVID-19 (coronavirus disease of 2019) induced ARDS (acute respiratory distress syndrome). The patients will be assigned in a 1:1 ratio to receive standard treatment protocol plus inhaled Low molecular weight heparin. The primary objective is to determine the hypoxemia improvement on a 5-point clinical scale for COVID-19 induced ARDS patients.

DETAILED DESCRIPTION:
Lungs are the major target organ of COVID-19, caused by the SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2). Multiple drug options have been evaluated for efficacy against worsening symptoms of COVID-19 patients. Low molecular weight heparin, known for its antiviral and anti-inflammatory effect, was determined to be applicable for ARDS-induced Hypoxemia.

In cases of viral diseases that primarily targets the lungs, oral drugs and parenteral applications have shown to be insufficient due to low drug accumulation in the target organ site. An increase in drug dosage in order to achieve the necessary drug concentration leaves the patient with intolerable side effects. An inhalation delivery route of the drug would not only directly target the lungs but would also require less dosage. This is expected to increase patient tolerability and the efficacy of the treatment.

Soft mist inhalers are advantageous above the other inhalation devices, for it reaches a higher retention rate in the lungs. Furthermore, the device to be used in this clinical study provides an "enclosed system" which decreases the risk of environmental contamination, thus is meant to protect healthcare professionals or to minimize associated contamination risks.

This Phase-IIb clinical trial is to include 40 critically ill COVID-19 induced ARDS patients, that will receive Low molecular Weight Heparin via a soft mist inhaler at a dose of 4000 IU per administration, twice a day for 10 days in addition to the standard treatment determined by the Turkish Ministry of Health. A total of 80 patients will be enrolled, in which the drug receiving group will be assigned. The primary outcome of the clinical study is the improvement of ARDS induced hypoxemia on a 5-scale determination method at the end of the 10th day. The study inquires to perceive the early effects of inhaled Low molecular weight heparin on critically ill COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* Positive reserve transcriptase polymerase chain reaction (RT-PCR) test of nasopharyngeal swab for COVID- 19, and pneumonia confirmed by a Computed Tomography (CT).
* Negative reserve transcriptase polymerase chain reaction (RT-PCR) test of nasopharyngeal swab for COVID- 19, but radiological and biochemical examinations unambiguously suggest COVID-19, when other possible diagnoses were excluded.

Exclusion Criteria:

* Pregnancy
* History of heparin and associated drug allergies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-05-21 (Actual)

PRIMARY OUTCOMES:
Change in clinical status on a 5-point clinical scale for hypoxemia | Days 1-10
  * Level 1: if the patient can breathe comfortably in the room air.
  * Level 2: if the peripheral oxygen saturation improves with an oxygen therapy up to 6 L/min via nasal cannula.
  * Level 3: If it can be improved with a 500 mL reservoir oxygen mask with 15 L/min oxygen treatment.
  * Level 4: If it can be improved with high flow oxygen therapy.
  * Level 5: If the intubation is the only choice.

SECONDARY OUTCOMES:
Improvement rate of the breathing status | Day 1 and Day 10
  Change in number of patients that were able to breath in room air will be compared on Day 1 and Day 10 (Comparison between the Treatment Group and Control Group)
Change in peripheral oxygen saturation (Sp02) | Days 1-10
  A change in SpO2 levels in the duration of the study (SpO2 < % 95)
Length of stay | Days 1-10
  Number of patients administered to intensive care unit (ICU)
Overall survival | Days 1-10
  During or post-study follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Ayca Yildiz-Pekoz, PhD, Study Chair — Istanbul University Faculty of Pharmacy; Mustafa Erelel, MD, Study Director — Istanbul University Faculty of Medicine
Locations (1):
- Istanbul University Medical Faculty, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data sharing will be decided on a later date depending on completion of further study Phases

REFERENCES:
- See also: Republic of Turkey Ministry of Health website on COVID-19 — http://covid19.saglik.gov.tr